CLINICAL TRIAL: NCT04016441
Title: Cost and Quality in Consumer Sunscreen Preferences
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: RVK06052019
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: sunscreen
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Subjects who are capable of completing an online, English survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will complete a survey online

SUMMARY:
This study seeks to determine what price consumers are willing to pay for a sunscreen product containing their ideal combination of attributes or qualities. This study will assess consumer preferences for various sunscreen qualities, as well as the relative contribution of each preference to the consumer's monetary valuation of a complete sunscreen product. The hypothesis is that respondents' willingness to pay for each sunscreen attribute will vary by demographic characteristics, especially self-identified race and socioeconomic class

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 years old or older.
* Subjects who are capable of completing an online, English survey.

Exclusion Criteria:

* Subjects less than 18 years old
* Subjects who have previously completed the study.
* Subjects who are not able to complete an online, English survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is a cross-sectional study of self-identified sunscreen users age 18 years and older.
Sampling Method: Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of sunscreen preference differences between ideal and willingness to pay | 1 year
  The frequency at which research participants indicate ideal sunscreen preferences versus willingness to pay for such preferences will be assessed in the questionnaire. The unit of measure will be a numerical value, number of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States